CLINICAL TRIAL: NCT02358070
Title: Epidemiologic Study of Hepatocellular Carcinoma in the US
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: HEP0049
Record Dates: First submitted 2015-01-29; First posted 2015-02-06 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — saliva samples

GROUPS / COHORTS (2):
- HCC group
- control group

SUMMARY:
The purpose of this study is:

* to investigate the risk factors of HCC among Americans with focus on lifestyle factors and energy balance.
* to identify single nucleotide polymorphisms (SNPs) and haplotypes that are associated with HCC risk through a genome-wide search.
* to assess if genetic susceptibility differs by hepatitis virus infection or lifestyle factors, and to explore if there are interplays or effect modifications between genetic factors and viral infection or lifestyle factors.

ELIGIBILITY:
Inclusion Criteria for HCC cases:

* a diagnosis of primary liver cancer (excluding secondary tumors)
* a diagnosis of hepatocellular carcinoma if histology is available (excluding those diagnosed in intrahepatic bile duct, bile canals, biliary passages, canaliculi, gall duct and gallbladder)
* a diagnosis of hepatocellular carcinoma with or without microscopic evaluation (including those diagnosed with clinical evidence, lab tests and direct visualization or radiographic and other imaging evidence)
* a histology of primary hepatocellular carcinoma when the patients had a prior diagnosis of other forms of cancer (excluding those who had no histological diagnosis of hepatocellular carcinoma while having a prior history of other cancer;
* age at diagnosis between 35 and 84 years
* living in Connecticut, New Jersey, New York, or Hawaii for at least a year as regular residents.

Exclusion Criteria for HCC cases:

* uncertain diagnoses or classification of malignancy, such as unknown origin
* a diagnosis of primary tumors in other organs, not in the liver
* unable to communicate well enough in English or Spanish
* having medical conditions, such as mental disorders, that prevent the subject from providing reasonably comprehensible information or from being able to give informed consent.
* diagnosed at age <35 years or >84 years
* temporary residents of New Jersey, Connecticut, New York, or Hawaii

Inclusion Criteria for control subjects:

* age between 35 and 84 years
* living in New Jersey or Connecticut for at least a year as regular residents
* able to communicate well in English or Spanish
* having no medical conditions, such as mental disorders, that prevent them from providing adequately comprehensible information
* potential subjects with a previous history of cancer are eligible.

Exclusion Criteria for control subjects:

* age < 35 years or > 84 years
* temporary residents of New Jersey or Connecticut
* unable to speak English or Spanish
* cannot provide adequately comprehensible information

Ages: 35 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with Hepatocellular Carcinoma in New Jersey and Connecticut as well as selected patients in New York, Hawaii and northern California.
  Healthy volunteers will comprise a random sample of New Jersey and Connecticut residents as controls.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
Lifetime physical activity | 20 years
  Lifetime physical activity will be measured by collecting data on major types of physical activity separately and by determining frequency, intensity, and duration of each activity using a combined modification of Friedenreich's lifetime physical activity questionnaire and Kriska's past year physical activity questionnaires.
Energy intake | 20 years
  A modified Food Frequency questionnaire based on one developed by Dr. Alan Kristal from the Fred Hutchinson Cancer Research Center (FHCRC) in Seattle will capture energy intake by differentiating low-fat food options from higher-fat counterparts.
Lifestyle factors | 20 years
  Structured questionnaires will be used to elicit information on demographic, anthropometric, and socioeconomic factors, long-term use of medications, medical history, and family history of cancer, cigarette smoking and alcohol consumption, physical activity, and dietary habits. Additional information unrelated to liver cancer will be included in the questionnaire to help assess possible recall bias.

CONTACTS AND LOCATIONS:
Overall Officials: Mindie Nguyen, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Liver Transplant Clinic, Stanford, California, United States